CLINICAL TRIAL: NCT03740321
Title: Superior Rectal Artery Embolization With Tri-acryl Gelatin Particles for Treatment of Symptomatic Hemorrhoids: Safety and Efficacy
Brief Title: SRAE With Embospheres for Hemorrhoids.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fahrettin Kucukay,MD, Prof.Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 80558721/237
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Embolization; Hemorrhoids
Keywords: Hemorrhoids; Superior rectal artery; embolization; microspheric particles
MeSH Terms: conditions — Hemorrhoids | interventions — Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: Blocked randomized, single blind, prospective study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Embospheres 500-700 microns (Experimental): Intervention.Embolization with 500-700 micron particles will be performed with 1 ml vials. Embolization procedure will be continued with vials until the stasis in SRAE will be achieved. Procedure will be performed only one time.
  Interventions: Device: Embolization with tri-acryl gelatin (Embosphere) particles
- Embospheres 700-900 microns (Experimental): Intervention.Embolization with 700-900 micron particles will be performed with 1 ml vials. Embolization procedure will be continued with vials until the stasis in SRAE will be achieved. Procedure will be performed only one time.
  Interventions: Device: Embolization with tri-acryl gelatin (Embosphere) particles

INTERVENTIONS:
Device: Embolization with tri-acryl gelatin (Embosphere) particles — Left, right and posterior branches of superior rectal artery will be embolized with tri-acryl gelatin particles in 500-700 and 700-900 micrometers in size until homeostasis will be achieved.
  Other Names: Embosphere

SUMMARY:
In this study , safety and efficacy of superior rectal artery embolization with embospheres will be researched prospectively.

DETAILED DESCRIPTION:
Symptomatic hemorrhoidal disease is a still important public health problem although there are many surgical and nonsurgical minimal invasive treatment methods. Treatment methods are not satisfactory or invasive in some percent of the patients. Superior rectal artery embolization(SRAE) for hemorrhoids is an adapted technique derived from Doppler-guided hemorrhoidal artery ligation (DGHAL). In this technique, the distal branches of the superior rectal artery arising from the inferior mesenteric artery is occluded endovascularly with coils. Its feasibility and safety were supported by articles. Collateralization and recurrence was seen following coil embolization. To prevent this , tri-acryl gelatin microspheres in 500-700 and 700-900 micrometers in size will be used. Safety and efficacy of embolization and using different sized particles will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of hemorrhoidal disease
* Patients with written informed consent
* Patients refusing surgery or other interventional methods
* Patients with high risk for surgery
* Patients accepting follow ups

Exclusion Criteria:

* Previous intervention
* Colorectal diseases other than hemorrhoids
* Patients with anal stenosis
* Patients with rectal prolapsus
* pregnant patients
* Patients with contraindications for technical steps or contrast usage.
* Patients do nor or could not give written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure related mortality (safety) | 12 month
  The mortality rate among the patients during 12 months related with interventional procedure.
Incidence of procedure related complications (safety) | 12 month
  The morbidity rate among the patients during 12 months related with interventional procedure.
Incidence of the patients' being free of symptoms from hemorrhoidal disease (efficacy) | 12 month
  The efficacy and clinical success of the procedure will be evaluated

SECONDARY OUTCOMES:
Technical success | On the day of intervention
  The rate of interventions that were performed successfully.
Recurrence | 3-6-12. months
  Recanalization or collateralization of the previously embolized rectal arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Fahrettin Kucukay, Study Chair — Eskisehir Osmangazi University, Faculty of Medicine, Department of Interventional Radiology
Locations (1):
- Eskisehir Osmangazi University, Faculty of Medicine, Department of Interventional Radiology, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zakharchenko A, Kaitoukov Y, Vinnik Y, Tradi F, Sapoval M, Sielezneff I, Galkin E, Vidal V. Safety and efficacy of superior rectal artery embolization with particles and metallic coils for the treatment of hemorrhoids (Emborrhoid technique). Diagn Interv Imaging. 2016 Nov;97(11):1079-1084. doi: 10.1016/j.diii.2016.08.002. Epub 2016 Aug 31. PMID 27597728
- [Result] Vidal V, Sapoval M, Sielezneff Y, De Parades V, Tradi F, Louis G, Bartoli JM, Pellerin O. Emborrhoid: a new concept for the treatment of hemorrhoids with arterial embolization: the first 14 cases. Cardiovasc Intervent Radiol. 2015 Feb;38(1):72-8. doi: 10.1007/s00270-014-1017-8. Epub 2014 Nov 4. PMID 25366092
- [Result] Vidal V, Louis G, Bartoli JM, Sielezneff I. Embolization of the hemorrhoidal arteries (the emborrhoid technique): a new concept and challenge for interventional radiology. Diagn Interv Imaging. 2014 Mar;95(3):307-15. doi: 10.1016/j.diii.2014.01.016. Epub 2014 Feb 28. PMID 24589187
- [Result] Galkin E. [X-ray endovascular embolization of the superior rectal artery: New potentialities in the surgical management of chronic hemorrhoids]. Vestn Rentgenol Radiol. 2001 Nov-Dec;(6):44-9. Russian. PMID 11858033
- [Result] Tradi F, Louis G, Giorgi R, Mege D, Bartoli JM, Sielezneff I, Vidal V. Embolization of the Superior Rectal Arteries for Hemorrhoidal Disease: Prospective Results in 25 Patients. J Vasc Interv Radiol. 2018 Jun;29(6):884-892.e1. doi: 10.1016/j.jvir.2018.01.778. Epub 2018 Apr 30. PMID 29724519
- [Result] Venturini M, De Nardi P, Marra P, Panzeri M, Brembilla G, Morelli F, Melchiorre F, De Cobelli F, Del Maschio A. Embolization of superior rectal arteries for transfusion dependent haemorrhoidal bleeding in severely cardiopathic patients: a new field of application of the "emborrhoid" technique. Tech Coloproctol. 2018 Jun;22(6):453-455. doi: 10.1007/s10151-018-1802-5. Epub 2018 May 24. No abstract available. PMID 29797246
- [Result] Primo Romaguera V, Gregorio Hernandez A, Andreo Hernandez L, de la Morena Valenzuela E. Selective embolization of the superior rectal artery: An alternative to hemorrhoid surgery? Cir Esp (Engl Ed). 2018 Apr;96(4):239-241. doi: 10.1016/j.ciresp.2017.08.005. Epub 2017 Oct 14. No abstract available. English, Spanish. PMID 29042023
- See also: Device descriptions, Instructions for use — https://www.merit.com/interventional-oncology-spine/embolotherapy/microspheres/embosphere-microspheres/

DOCUMENTS (1):
  • Study Protocol (2017-07-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03740321/Prot_000.pdf